CLINICAL TRIAL: NCT00004091
Title: Development of Antibody-Based Diagnostic Markers for Abnormal Cervical Cells
Brief Title: Detection of Biomarkers in Abnormal Cervical Cells in Women With Abnormal Pap Test Results
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: John Lurain, MD, Northwestern University
Other Study IDs: NU 99G3; NU-99G3; NCI-G99-1582
Record Dates: First submitted 1999-12-10; First posted 2004-03-01 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Cervical Cancer
Keywords: cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Papanicolaou Test; Fluorescent Antibody Technique

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

INTERVENTIONS:
Other: Papanicolaou test
Other: cytology specimen collection procedure
Other: fluorescent antibody technique
Procedure: colposcopic biopsy
Procedure: study of high risk factors

SUMMARY:
RATIONALE: Examining biomarkers in abnormal cervical cells may improve the ability to detect these cells and plan effective treatment.

PURPOSE: Diagnostic trial to detect specific biomarkers in abnormal cervical cells in women who have abnormal Pap test results.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the detection of transferrin receptor, epidermal growth factor receptor, and the MaTu-MN protein in exfoliated cervical epithelial cells from women with abnormal Pap test using fluorescent labeled antibody probe vs histology.

OUTLINE: Patients undergo a Pap test and a colposcopy. Cervical epithelial cells are collected from the most abnormal appearing lesion. Cells are examined for molecular markers using a fluorescent antibody test. The presence or absence of these markers is compared to results of the Pap test and the histology of the cells.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study within 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of abnormal Pap test, as indicated by one of the following: Atypical squamous cells of undetermined significance (ASCUS) Low grade squamous intraepithelial lesion (LGSIL) High grade squamous intraepithelial lesion (HGSIL) Visible lesion on cervix by colposcopy

PATIENT CHARACTERISTICS: Age: Any age Performance status: ECOG 0-4 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Pregnant or nursing women allowed

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: No prior pelvic irradiation Surgery: No prior total hysterectomy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients must have a diagnosis of an abnormal Pap test, performed as part of standard of care screening in the clinic. The patient's informed consent will be obtained during their initial interview with the clinic physician.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 1999-08; Primary Completion 2001-02 (Actual); Study Completion 2001-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Y. Roland, MD, Study Chair — Florida Gynecologic Oncology - Fort Myers
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States